CLINICAL TRIAL: NCT05089162
Title: Evaluation de la Congestion en Hospitalisation de Jour Pour un Bilan d'Insuffisance Cardiaque Chronique à Fraction d'éjection altérée ou modérément altérée CHF-COV Reduced (Chronic Heart Failure With Reduced Ejection Fraction - COngestion eValuation)
Brief Title: CHF-COV Reduced (Chronic Heart Failure With Reduced Ejection Fraction - COngestion eValuation)
Acronym: CHF-COVReduced
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pr. Nicolas GIRERD (Other)
Responsible Party: Sponsor-Investigator, Pr. Nicolas GIRERD, Principal Investigator, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020PI145-2
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-03

CONDITIONS: Chronic Heart Failure; Reduced Ventricular Ejection Fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with chronic HF with reduced ventricular ejection fraction coming for scheduled day (Experimental)
  Interventions: Procedure: Clinical examination centered on congestion; Procedure: Cardiac, pulmonary, peritoneal, jugular and renal Doppler ultrasounds; Procedure: Blood sample retrieved for biological assessment and biobanking; Other: Telephone follow-up; Behavioral: Kansas City Cardiomyopathy Questionnaire (KCCQ)

INTERVENTIONS:
Procedure: Clinical examination centered on congestion — Clinical examination centered on congestion (including the EVEREST, ASCEND and Ambrosy scores) will be performed during day hospitalization or consultation
Procedure: Cardiac, pulmonary, peritoneal, jugular and renal Doppler ultrasounds — Cardiac, pulmonary, peritoneal, jugular and renal Doppler ultrasounds and liver elastography will be performed during day hospitalization or consultation/ peritoneal, jugular and renal Doppler ultrasounds are optional
Procedure: Blood sample retrieved for biological assessment and biobanking — Blood sample retrieved for biological assessment and biobanking will be performed during day hospitalization or consultation
Other: Telephone follow-up — Telephone follow-up will be performed 3, 12 and 24 months after day hospitalization or consultation
Behavioral: Kansas City Cardiomyopathy Questionnaire (KCCQ) — Questionnaire centered on patient's quality of life at discharge and 3, 12 and 24 months after discharge

SUMMARY:
Heart failure (HF) is a significant cause of death and the leading cause of hospitalization in patients over 65 years of age. Congestion is the main source of symptoms and the leading cause of hospitalization for HF. Furthermore, congestive signs identified in asymptomatic patients are associated with the risk of developing symptomatic HF. The literature supports a multi-modality / integrative evaluation of congestion, combining clinical examination, laboratory results and ultrasound evaluation.

The main objective of the CHF-COVReduced study is to identify congestion markers (clinical, biological and ultrasound) quantified during a consultation or day hospitalization for the monitoring of chronic HF with reduced left ventricular ejection fraction that are associated with the risk of all-cause death, hospitalization for acute HF or IV diuretics injection in a day hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic acute heart failure with reduced ventricular ejection fraction admitted in hospital for scheduled day hospitalization or in consultation
* Patient with altered (left ventricular ejection fraction <40%) and moderately altered (left ventricular ejection fraction between 40 and 50%) left ventricular ejection fraction
* Age ≥18 years
* Patients having received complete information regarding the study design and having signed their informed consent form.
* Patient affiliated to or beneficiary of a social security scheme.

Exclusion Criteria:

* Comorbidity for which the life expectancy is ≤ 3 months
* Dialysis patient (peritoneal dialysis or hemodialysis) or patients with glomerular filtration rate <15 ml/min/m2 at inclusion.
* History of lobectomy or pneumonectomy lung surgery
* Severe pulmonary or pleural pathology preventing reliable acquisition of lung ultrasound images: severe emphysema, chronic pleurisy, pulmonary fibrosis, etc.
* Pregnant woman, parturient or nursing mother
* Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* Adult person who is unable to give consent
* Person deprived of liberty by a judicial or administrative decision,
* Person subject to psychiatric care pursuant to Articles L. 3212-1 and L. 3213-1 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2028-12-14 (Estimated); Study Completion 2029-06-14 (Estimated)

PRIMARY OUTCOMES:
Rate of death from all causes | 24 months after day hospitalization or consultation
  composite endpoint : rate of death from all causes, hospitalisation for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 2 and 3)
Rate of hospitalisation for acute heart failure | 24 months after day hospitalization or consultation
  composite endpoint : rate of death from all causes, hospitalisation for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 1 and 3)
Rate of day-hospital or in-home IV diuretics injection for acute HF | 24 months after day hospitalization or consultation
  composite endpoint : rate of death from all causes, hospitalisation for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 1 and 2)

SECONDARY OUTCOMES:
Rate of death from all causes | 24 months after day hospitalization or consultation
  composite endpoint of rate of death from all causes or hospitalisation for acute heart failure 24 months after day hospitalization (with outcome 5)
Rate of hospitalisation for acute heart failure | 24 months after day hospitalization or consultation
  composite endpoint of rate of death from all causes or hospitalisation for acute heart failure 24 months after day hospitalization (with outcome 4)
Rate of death from all causes | 24 months after day hospitalization or consultation
Rate of hospitalisation for acute heart failure | 24 months after day hospitalization or consultation
  composite endpoint: Rate of hospitalisation for acute heart failure or day-hospital/in-home IV diuretics injection for acute HF 24 months after day hospitalization (with outcome 8)
Rate of day-hospital or in-home IV diuretics injection for acute HF | 24 months after day hospitalization or consultation
  composite endpoint: Rate of hospitalisation for acute heart failure or day-hospital/in-home IV diuretics injection for acute HF 24 months after day hospitalization (with outcome 7)
Rate of hospitalisation for cardiovascular reason | 24 months after day hospitalization or consultation
Rate of death from all causes | 3, 12 and 24 months after day hospitalization or consulation
  composite endpoint: Rate of hospitalisation for acute heart failure or day-hospital/in-home IV diuretics injection for acute HF 24 months after day hospitalization (with outcome 11)
Rate of hospitalisation for acute heart failure | 24 months after day hospitalization or consultation
  composite endpoint: Rate of hospitalisation for acute heart failure or day-hospital/in-home IV diuretics injection for acute HF 24 months after day hospitalization (with outcome 10)
Rate of cardiovascular death | 24 months after day hospitalization or consultation
NYHA (New York Heart Association) class measured | 3, 12 and 24 months after day hospitalization or consultation
Natriuretic peptides | At inclusion
  BNP or Nt-Pro BNP
Renal function | At inclusion
  Assessed by glomerular filtration rate
Plasma volume | At inclusion
  calculated from haemoglobin and haematocrit value
Rate of Bilirubin | At inclusion
Rate of ASAT | At inclusion
Rate of ALAT | At inclusion
Rate of V factor | At inclusion
Blood potassium concentration | At inclusion
Circulating NtProBNP | At inclusion
Liver elastography value | At inclusion
  Measured with Fibroscan®
Quality of life assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) | At inclusion and 3, 6 and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No